CLINICAL TRIAL: NCT00982748
Title: Effects of Pranayama on Fatigue Among Patients Undergoing Chemotherapy
Brief Title: Yoga Breathing for Fatigue in Patients Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Anand Dhruva, Assistant Clinical Professor, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 08803; Mt.Zion Healthfund 20070658
Record Dates: First submitted 2009-09-18; First posted 2009-09-23 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: Fatigue; Chemotherapy; Yoga; Breathing; Cancer; Anxiety; Pranayama; Stress; Fatigue-associated symptoms in chemotherapy patients; Quality of life in chemotherapy patients
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Respiratory Aspiration; Neoplasms; Anxiety Disorders | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group B (Active Comparator): Study participants in this arm attend yoga breathing classes once per week over the span of one chemotherapy cycle.
  Interventions: Behavioral: Pranayama (Yoga Breathing) Techniques
- Group A (Experimental): Participants in this study arm attend weekly yoga breathing classes during two consecutive cycles of chemotherapy
  Interventions: Behavioral: Pranayama (Yoga Breathing) Techniques

INTERVENTIONS:
Behavioral: Pranayama (Yoga Breathing) Techniques — 1-hour long yoga breathing classes, taught once per week for 2-8 consecutive weeks. Dose (Number of classes) administered is dependent on randomization arm and individuals' chemotherapy cycle length.

SUMMARY:
The purpose of this study is to determine the feasibility and efficacy of yoga breathing techniques to manage fatigue and other cancer-related side effects, in cancer patients undergoing chemotherapy.

DETAILED DESCRIPTION:
Fatigue is the most common complaint among cancer patients. This pilot study will evaluate the effects of pranayama (ancient yoga breathing techniques) on fatigue and quality of life among 30 patients undergoing chemotherapy, on an every 2, 3, or 4 week schedule, with a fatigue score of at least 4 on a scale of 0 (none) to 10 (most). Patients will be randomized to either pranayama or wait-list control. The pranayama group will learn and practice 3 breathing techniques on a daily basis. The study period will occur during 2 consecutive cycles of chemotherapy (cycle A and Cycle B), and the wait-list control patients will crossover to the treatment arm at the beginning of his/her Cycle B. Fatigue will be measured using the revised Piper Fatigue Scale along with quality of life measures. These study measures will be conducted at baseline, at the end of cycle A, and at the end of cycle B. We hypothesize that pranayama will improve clinical symptoms of fatigue and quality of life among patients undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of cancer that requires at least 2 further cycles of chemotherapy on an every 14, 21, or 28 day schedule
* A score of at least 4/10 on a 0-10 (0-none, 10-most) visual analog scale for fatigue at the time of enrollment
* Able to read, write and understand English
* Karnofsky Performance Status greater than 60
* Ability to give informed consent

Exclusion Criteria:

* Severe COPD
* Receiving chronic oxygen therapy
* Congestive heart failure: NYHA class 3 or greater
* Transfusion dependent anemia
* Uncontrolled thyroid disease
* Advance kidney disease requiring dialysis
* Advance liver disease
* More than three previous chemotherapy regimens
* Current, ongoing yoga breathing practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Feasibility | Baseline and second cycle of chemotherapy
  Feasibility will be evaluated based on recruitment, retention, completion of study classes and home practice, and completion of study measures

SECONDARY OUTCOMES:
Cancer associated symptoms and quality of life | baseline and final cycle of chemotherapy
  fatigue, sleep, stress, anxiety and depression quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Osher Center for Integrative Medicine, UCSF, San Francisco, California, United States

REFERENCES:
- [Derived] Dhruva A, Miaskowski C, Abrams D, Acree M, Cooper B, Goodman S, Hecht FM. Yoga breathing for cancer chemotherapy-associated symptoms and quality of life: results of a pilot randomized controlled trial. J Altern Complement Med. 2012 May;18(5):473-9. doi: 10.1089/acm.2011.0555. Epub 2012 Apr 23. PMID 22525009